CLINICAL TRIAL: NCT02522039
Title: Effect of Topical Anti-glaucoma Medications on Late Pupillary Light Reflex, as Evaluated by Pupillometry
Brief Title: Pupillary Response After Glaucoma Medication
Acronym: pupil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Birgit Sander, md, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GlostrupUH
Record Dates: First submitted 2014-11-14; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Drug Effect (Glaucoma Drugs)
MeSH Terms: interventions — Latanoprost; Timolol; dorzolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Latanoprost (Experimental): solution, 1 drop of 50ug/ml latanoprost, was given to study eye after washout period of 1 week between drugs
  Interventions: Drug: Latanoprost
- Timolol (Experimental): solution, 1 drop of 5mg/ml timolol , was given to study eye after washout period of 1 week between drugs
  Interventions: Drug: Timolol
- dorzolamide (Experimental): solution, 1 drop of 20 mg/ml dorzolamide, was given to study eye after washout period of 1 week between drugs
  Interventions: Drug: Dorzolamide
- Other (No Intervention): no drug given and pupil measurements were performed before and at 30 and 180 min at equivalent hours as drugs measurements

INTERVENTIONS:
Drug: Latanoprost — 1 drop of latanoprost was given to study eye after washout period of 1 week between drugs
  Arms: Latanoprost
Drug: Timolol — 1 drop of timolol was given to study eye after washout period of 1 week between drugs
  Other Names: Optimol
  Arms: Timolol
Drug: Dorzolamide — 1 drop of dorzolamide was given to study eye after washout period of 1 week between drugs
  Arms: dorzolamide

SUMMARY:
Investigation of the effect on the pupillary constriction by latanoprost, dorzolamide,timolol in healthy subjects. The pupillary constriction is compared to no drug.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* ophthalmological diseases
* systemic disease
* smoking
* refractive error >= 6 diopters

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
pupillary constriction measured as the post-illimination pupillay response (PIPR) | 1 day
  The pupillary diameter 0 to 10 seconds after light stimulation, the diameter is measured relative to the initial dark adapted pupil diameter

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Lund-Andersen, Professor, Study Director — Head of the project
Locations (1):
- Glostrup University Hospital, Glostrup Municipality, Denmark